CLINICAL TRIAL: NCT07029789
Title: Clinical Evaluation of Deep Learning-Enhanced Super-Resolution Single-Beat CMR: Prospective Comparison Study
Brief Title: Deep Learning Super-Resolution Single-Beat CMR
Acronym: DL-SB-CMR
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Isaak, Radiologist, Radiology Clinic, University Hospital, Bonn
Other Study IDs: 2024-379-BO
Record Dates: First submitted 2025-06-03; First posted 2025-06-19 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Heart Diseases; Myocardial Disease
Keywords: deep learning; cardiovascular magnetic resonance; image reconstructions; cardiac imaging techniques; single-beat; super-resolution; accelerated imaging
MeSH Terms: conditions — Heart Diseases; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient cohort: * suspected myocardial disease with clinical indication for CMR
  * undergoing one CMR with two integrated protocols (standard and DL single beat protocol)

SUMMARY:
Deep learning super-resolution reconstruction is an emerging technique that enhances the resolution of cardiac magnetic resonance (CMR) scans beyond the original acquisition through post-processing. This study investigates whether a deep learning-based single-beat super-resolution CMR protocol-including cine, T2-STIR, and LGE sequences-can provide diagnostic equivalence to a standard segmented CMR protocol. Total scan time, diagnostic confidence, and diagnostic interchangeability are compared between protocols, with particular focus on wall motion abnormalities, myocardial edema, pericardial effusion, late gadolinium enhancement and final diagnosis. The goal is to assess diagnostic interchangeability while improving efficiency and motion robustness.

DETAILED DESCRIPTION:
Cardiac magnetic resonance (CMR) is the gold standard for non-invasive assessment of myocardial diseases, providing comprehensive information through e.g. cine imaging, T2-weighted sequences, and late gadolinium enhancement (LGE). Conventional CMR protocols typically rely on segmented (multi-shot) acquisitions over multiple heartbeats and require repeated breath-holds, which can limit patient comfort and compliance. While these segmented sequences offer high spatial resolution, they are prone to motion and respiratory artifacts-particularly in patients with arrhythmias or dyspnea-and contribute to long total examination times.

Recent advances in deep learning (DL) reconstruction techniques have enabled substantial acceleration of segmented CMR sequences, particularly for cine and LGE imaging. These approaches effectively reduce acquisition time but still rely on regular cardiac rhythm and adequate breath-holding capacity, limiting their applicability in more challenging patient populations. In contrast, single beat (or: single-shot) imaging acquires data within a single heartbeat, offering a motion-robust alternative, though at the cost of lower spatial resolution.

Efforts to streamline CMR are ongoing, with some studies proposing to reduce comprehensive exam times to 30 minutes or less. In parallel, full DL-based reconstruction MRI protocols are being increasingly explored across MRI domains, including neuroimaging and musculoskeletal imaging. Applying deep learning super-resolution to CMR, particularly in combination with single-beat acquisitions with the option of free-breathing acquisition, may enhance both speed and robustness.

This prospective investigates whether a deep learning-based single-beat super-resolution CMR protocol - including single-shot cine, T2-STIR, and LGE sequences in both short- and long-axis views - can provide diagnostic interchangeability to a standard segmented protocol. All participants undergo both protocols during the same exam session. Total scan times are compared between protocols using Student's t-test. Three blinded readers evaluate predefined diagnostic categories including wall motion abnormalities, pericardial effusion, myocardial edema, LGE, and the final CMR diagnosis. Generalized estimating equations with bootstrapped 95% confidence intervals and a predefined equivalence margin of ±5% was used for the interchangeability analysis. Agreement in categorical ratings was evaluated using Cohen's Kappa and Fleiss' Kappa, as appropriate. Diagnostic confidence was rated on a 5-point Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for CMR
* Aged 18 years or older.
* Willing to participate in the study.
* Able and willing to provide signed informed consent.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Non-removable magnetic metallic implants, prosthetic devices, or extensive tattoos covering large areas of the body
* Presence of a non-MRI safe pacemaker or neurostimulator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical indication for CMR
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic interchangeability | May - December 2024
  Assessment of diagnostic interchangeability between the deep learning-based single-beat SuperRes CMR protocol and the standard segmented CMR protocol. Diagnostic categories include wall motion abnormalities, pericardial effusion, myocardial edema, late gadolinium enhancement, and the final CMR diagnosis. Interchangeability was evaluated using generalized estimating equations with bootstrapped 95% confidence intervals and a predefined equivalence margin of ±5%. For each category, the outcome is expressed as an individual equivalence index (%), defined as the difference in agreement probabilities.

SECONDARY OUTCOMES:
Scan time | May - December 2024
  Comparison of total scan duration between the deep learning-based single-beat SuperRes CMR protocol and the standard segmented CMR protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Isaak, PD Dr., Principal Investigator — University Hospital Bonn, Germany; Julian Luetkens, Prof., Study Director — University Hospital Bonn, Germany
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided